CLINICAL TRIAL: NCT05554991
Title: Efficacy and Tolerability of a Composition Comprising of HMO in a Supplement Format on Colic Management: a Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Human Milk Oligosaccharide (HMO) Supplementation in Colic Management
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Impossibility to recruit the targeted population
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20.28.INF
Record Dates: First submitted 2022-03-28; First posted 2022-09-26 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Colic
MeSH Terms: conditions — Colic | interventions — Health Maintenance Organizations; Palliative Care

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled, parallel-arm, intervention study
Who Masked: Participant, Investigator
Masking Description: Randomization will be carried out using iMedidata Randomization Trial Supply Management System with the dynamic allocation algorithm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liquid oral supplement comprising HMO (Experimental): 2 ampules/day for 21 days
  Interventions: Dietary Supplement: HMO; Behavioral: Parental reassurance and support
- Placebo (Placebo Comparator): 2 ampules/day for 21 days
  Interventions: Dietary Supplement: Placebo; Behavioral: Parental reassurance and support

INTERVENTIONS:
Dietary Supplement: HMO — Composition comprising of HMO
  Arms: Liquid oral supplement comprising HMO
Dietary Supplement: Placebo — Placebo supplementation having the same appearance and dosing regimen as the intervention
  Arms: Placebo
Behavioral: Parental reassurance and support — Both groups will receive standardized written materials to provide parental reassurance and support, in alignment with local clinical practice

SUMMARY:
Efficacy and tolerability of a composition comprising of HMO in a supplement format on colic management: a double-blind, randomized, placebo-controlled trial

DETAILED DESCRIPTION:
This is a double-blinded, randomized, placebo-controlled trial. The purpose of this trial is to investigate the efficacy and tolerability of a composition comprising of HMO in a supplement format in the management of colicky infants aged 2-12 weeks.

ELIGIBILITY:
Inclusion criteria:

1. Infants 2 weeks - 12 weeks of age at enrolment
2. Infants diagnosed with colic according to Rome IV criteria: Diagnostic criteria for research purposes (infant must meet all Rome IV criteria):

   1. An infant who is less than 5 months of age (in the current clinical trial, only infants 2 weeks to 8 weeks of age will be enrolled) when the symptoms start and stop
   2. Recurrent and prolonged periods of infant crying, fussing, or irritability reported by caregivers that occur without obvious cause and cannot be prevented or resolved by caregivers
   3. No evidence of infant failure to thrive, fever, or illness
   4. Excessive crying/fussiness for 3 or more hours per day during 3 or more days in the past 7 days as reported by parents to the clinician
   5. Total 24-hour crying plus fussing is 3 hours or more when measured by at least one prospectively kept 24-hour behavior diary. (The Structured Infant Crying and Fussing Diary will be dispensed at the screening visit (V0), completed for two 24-hour periods at H0 (days -3 to -1), and returned at V1 to be used as part of the diagnostic criteria for infantile colic.)
3. Term infants (≥ 37 weeks) generally healthy with normal birth weight (≥2.5kg) and singleton born
4. Predominantly formula fed* (formula fed ≥ 80% of the time) for at least 7 days before randomization and the choice of formula feeding has been made by the parents before the beginning of the trial.
5. Infants who have been on the same formula for the past 5 days
6. Signed informed consent obtained for infant's and parents'/Legally Acceptable Representative (LAR) participation in the study
7. Parent/LAR of infant agrees not to enroll infant in another interventional clinical research study while participating in this study
8. Parent of the infant/LAR is willing and able to fulfill the requirements of the study protocol
9. Parent of infant can be contacted throughout the study

   * Predominantly formula feeding defined in the study means that the infant's predominant source of nourishment is formula. Specifically, infants are fed with formula for at least 80% of total milk feeds per day.

Exclusion criteria:

1. Presence of any congenital condition and/or previous or current illness/infection and (or) medication use that could interfere with the main study outcomes.
2. Clinical evidence of chronic illness or gastrointestinal disorders, major medical problems (e.g. ill, immunocompromised, major developmental or genetic abnormality).
3. Known cow's milk protein allergy, lactose intolerance, or galactosaemia; including presence of any allergic manifestations.
4. Received any special formula (e.g. lactose-free, hydrolyzed protein) within 5 days before randomization or switched formulas within 5 days before randomization.
5. Received any of the following products/medication within 5 days before randomization:

   * Antibiotics
   * Alginate
   * Prokinetics
   * Proton pump inhibitors
   * Simethicone
   * L. reuteri probiotic
   * Formula containing Human milk Oligosaccharides
6. Other infant(s) <6months of age living in the same household.
7. Current participation in another interventional clinical trial.

Ages: 2 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Difference in average infant daily crying and fussing duration | At the end of the intervention period (day 21)
  Difference in average infant daily crying and fussing duration at the end of the intervention in the Intervention Group (IG) versus the Control Group (CG). The crying and fussing duration is measured using a structured infant crying and fussing diary.

SECONDARY OUTCOMES:
Modulation of infant gut microbiota (communities of microbes, their taxonomy, strain composition, diversity, ecology, functionalities, and the metabolites produced) | V1 (day 0), V2 (day 7), and V4 (day 21)
  Modulation of infant gut microbiota in the intervention group versus the control group assessed using metagenomics
Difference in average infant daily crying duration | Change from baseline (V1) to intervention end (V4)
  Difference in average infant daily crying duration at the end of the intervention in the IG versus the CG assessed using a structured infant crying and fussing diary.
Difference in average infant daily fussing duration | Change from baseline (V1) to intervention end (V4)
  Difference in average infant daily fussing duration at the end of the intervention in the IG versus the CG assessed using a structured infant crying and fussing diary.
Difference in average infant daily crying and fussing duration in the IG | Change from baseline (V1) to intervention end (V4)
  Difference in average infant daily crying duration and fussing duration combined from baseline (V1) to intervention end (V4) in the IG assessed using a structured infant crying and fussing diary.
Difference in average infant daily crying duration in the Intervention group | Change from baseline (V1) to intervention end (V4)
  Difference in average infant daily crying duration from baseline (V1) to intervention end (V4) in the Intervention group assessed using a structured infant crying and fussing diary.
Difference in average infant daily fussing duration in the Intervention group | Change from baseline (V1) to intervention end (V4)
  Difference in average infant daily fussing duration from baseline (V1) to intervention end (V4) in the interventional group assessed using a structured infant crying and fussing diary.
Infant daily crying and fussing duration assessed longitudinally | Longitudinal changes across specific visits V1 (day 0), V2 (day 7), V3 (day 14) and V4 (day 21)
  Infant daily crying and fussing duration combined assessed longitudinally across the intervention assessed using a structured infant crying and fussing diary.
Infant crying/fussing per 24 hours | At specific visits V1 (day 0), V2 (day 7), V3 (day 14) and V4 (day 21)
  Episodes of infant crying/fussing per 24 hours assessed using a structured infant crying and fussing diary.
Percentage of children achieving a reduction in daily crying and fussing | At specific visits V1 (day 0), V2 (day 7), V3 (day 14) and V4 (day 21)
  Percentage of children achieving a reduction in daily crying, fussing, crying and fussing time combined of ≤ 25 % and ≤ 50 % assessed using a structured infant crying and fussing diary.
Incidence of infantile colic | At specific visits V1 (day 0), V2 (day 7), V3 (day 14) and V4 (day 21)
  Incidence of infantile colic assessed using a structured infant crying and fussing diary.
Parental perception of colic severity | At specific visits V1 (day 0), V2 (day 7), V3 (day 14) and V4 (day 21)
  Parental perception of colic severity assessed using a 10-cm visual analog scale (VAS)
Overall GI tolerance and individual GI symptoms | V1 (day 0), V2 (day 7), V3 (day 14) and V4 (day 21)
  Overall infant GI tolerance and individual GI and GI-related symptoms (stooling, spitup/ vomiting, gassiness, crying, fussiness) assessed using IGSQ-13
Overall GI tolerance and individual GI symptoms | Baseline to intervention end (day 21)
  Change in IGSQ-13 scores assessed using IGSQ-13
Overall GI tolerance and individual GI symptoms | At V1 (day 0), V2 (day 7), V3 (day 14) and V4 (day 21)
  Functional GI symptoms (regurgitation, consistency of stools), crying, allergic symptoms (atopic eczema) and respiratory symptoms assessed using CoMiSS
Overall GI tolerance and individual GI symptoms | From baseline to intervention end (day 21)
  Change in CoMiSS scores assessed using CoMiSS
Overall GI tolerance and individual GI symptoms | 1-day retrospective GI diary at V1 (day 0) and prospective 3-Day GI symptom diary diaries at home (H2, H3 and H4) just prior to V2 (day 7), V3 (day 14) and V4 (day 21)
  Stool consistency, spitting up/vomiting and flatulence assessed using 1-day retrospective GI diary at V1 (day 0) and prospective 3-Day GI symptom diary diaries at home (H2, H3 and H4) just prior to V2 (day 7), V3 (day 14) and V4 (day 21)
Infant sleep | V1 (day 0), V2 (day 7), V3 (day 14) and V4 (day 21)
  Infant sleep duration and nighttime wakings per 24 hours assessed using Brief infant sleep questionnaire (BISQ)
Infant Quality of life | V1 (day 0), V2 (day 7), V3 (day 14) and V4 (day 21)
  Infant quality of life assessed using an Infant Quality of Life instrument. The tool includes IQI includes questions on 7 health items such as sleeping, crying, feeding , skin, breathing, playfulness and Interaction, and stooling. Each item consists of 4 levels, most of which are ranked by severity.
Parental and family quality of life | V1 (day 0), V2 (day 7), V3 (day 14) and V4 (day 21)
  Parental/family quality of life will be assessed using a Quality of Life Visual Analog Scale that rates the parent / family's quality of life based on a 10-point Likert scale.
Infant fecal gut microbiota | V1 (day 0), V2 (day 7), and V4 (day 21)
  Microbiome of fecal samples to investigate the communities of microbes, their taxonomy, strain composition, diversity, ecology, functionalities, and the metabolites produced assessed using metagenomics.
Fecal metabolism | V1 (day 0), V2 (day 7), and V4 (day 21)
  Fecal metabolism (pH, organic acids)
Fecal markers of inflammation calprotectin | V1 (day 0) and V4 (day 21)
  Inflammation biomarkers calprotectin assessed using ELISA.
Fecal markers of inflammation lipocalin | V1 (day 0) and V4 (day 21)
  Inflammation biomarkers lipocalin assessed using ELISA.
Infant anthropometry weight | V1 (day 0), V2 (day 7), V3 (day 14) (optional if V3 is a phone call) and V4 (day 21)
  Weight in grams
Infant anthropometry length | V1 (day 0), V2 (day 7), V3 (day 14) (optional if V3 is a phone call) and V4 (day 21)
  Length in cm
Infant anthropometry head circumference | V1 (day 0), V2 (day 7), V3 (day 14) (optional if V3 is a phone call) and V4 (day 21)
  Head circumference in cm
Infant anthropometry weight gain | V1 (day 0), V2 (day 7), V3 (day 14) (optional if V3 is a phone call) and V4 (day 21)
  Weight gain in g/d
Infant anthropometry length gain | V1 (day 0), V2 (day 7), V3 (day 14) (optional if V3 is a phone call) and V4 (day 21)
  Length gain in cm/d
Infant illness and infection and medication usage | V1 (day 0) until V4 (day 21)
  Data collected using a calendar-based electronic Infant Illness Diary (IID)

OTHER OUTCOMES:
Duration and number of episodes of infant crying type based on a crying-type classification of the audio recording | 24 hours after V1 (day 0), V2 (day 7), V3 (day 14) and for 3 days prior to V4 (day 21)
  Duration and number of episodes of each infant crying type (pain, fussiness, hunger) based on a crying-type classification of the audio recording
Proportion of children with a specific crying type based on a crying-type classification of the audio recording | 24 hours after V1 (day 0), V2 (day 7), V3 (day 14) and for 3 days prior to V4 (day 21)
  Proportion of children with a specific crying type (pain, fussiness, hunger) based on a crying-type classification of the audio recording
Duration of crying based on a crying-type classification of the audio recording | 24 hours after V1 (day 0), V2 (day 7), V3 (day 14) and for 3 days prior to V4 (day 21)
  Duration of crying based on a crying-type classification of the audio recording
Duration of fussing based on a crying-type classification of the audio recording | 24 hours after V1 (day 0), V2 (day 7), V3 (day 14) and for 3 days prior to V4 (day 21)
  Duration of fussing based on a crying-type classification of the audio recording
Duration of crying and fussing combined based on a crying-type classification of the audio recording | 24 hours after V1 (day 0), V2 (day 7), V3 (day 14) and for 3 days prior to V4 (day 21)
  Duration of crying and fussing combined based on a crying-type classification of the audio recording
Crying and fussing comparison between the structured infant crying and fussing diary and the crying-type classification of the recording of infant crying/fussing across the intervention | V1 (day 0), V2 (day 7), V3 (day 14) and V4 (day 21)
  Infant daily crying and fussing duration compared between the structured infant crying and fussing diary and the crying-type classification of the recording of infant crying/fussing across the intervention
Maternal Postpartum depression/ anxiety | V1 (day 0) and V4 (day 21)
  Maternal postpartum depressive and anxiety symptoms assessed using an Edinburgh postnatal depression scale (EPDS)

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (4):
  - Ospedale Pediatrico Giovanni XXIII, Policlinico di Bari, Bari
  - ASST FBF Sacco, Milan
  - AOUP Paolo Giaccone, Palermo
  - Azienda Ospedaliero -Universitaria Pisana, Pisa
- Spain (3):
  - Centro de Salud El Ranero, Murcia
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Unidad de Estudios e Investigación IHP, Seville

IPD SHARING:
Plan to Share IPD: No